Date: 2022 August 27

## COMPARISON OF ERECTOR SPINAE PLANE BLOCK WITH TRANSVERSUS ABDOMINIS PLANE BLOCK FOR POSTOPERATIVE PAIN MANAGEMENT IN PATIENTS UNDERGOING TOTAL ABDOMINAL HYSTERECTOMY: A RANDOMIZED CONTROLLED TRIAL

Biplov Neupane, Subash Prashad Acharya, Megha koirala, Basu dev Parajuli

## **INFORMED CONSENT FORM**

COMPARATIVE STUDY OF ERECTOR SPINAE PLANE BLOCK WITH TRANSVERSUS ABDOMINIS PLANE BLOCK FOR POSTOPERATIVE PAIN MANAGEMENT IN PATIENTS APPEARING FOR TOTAL ABDOMINAL HYSTERECTOMY

| | Department of | |
|---|---|---|
| M | Maharajgunj Medical Campus, Tribhuvan Unive<br>Maharajgunj, Katl | |
| I hav | e read and understood the information sheet ar | emale of years age, hereby confirm that ad consent form for this research being conducted ave had the opportunity to ask questions about it. |
| I here | eby declare that, | |
| | I understand that my participation in the study is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | |
| pe<br>th<br>He | I understand that the researchers, the IRC and other regulatory authorities will not need my permission to look at my health records both in respect of the current study and any further research that may be conducted in relation to it, even if I withdraw from the trial. I agree to this access. However, I understand that my identity will not be revealed in any information that will be published or released to the third parties. | |
| | I agree not to restrict the use of any data or results that arise from this study provided that such use is only for scientific purpose(s). | |
| 4. I a | agree to take part in this study. | |
| | ature (or Thumb impression) of the<br>arch participant/Legal Guardian | Signature (or Thumb impression) of Witness |
| Name | ature :e : | Signature: Name: Date: |
| Inves | stigator's | |
| Signa | ature: | |
| Name | e: | |
| Date | : | |